CLINICAL TRIAL: NCT01305161
Title: Diagnostic Accuracy of Flow Cytometry Applied to the Diagnosis of Peri-anaesthesic Reactions Induced by Neuromuscular Blockers
Brief Title: Flow Cytometry Applied to the Diagnosis of Peri-anaesthesic Reactions
Acronym: CYPREANE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Limoges (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: I09010
Record Dates: First submitted 2011-02-24; First posted 2011-02-28 (Estimated); Last update posted 2025-07-16 (Actual); Status verified 2019-01

CONDITIONS: Allergy
Keywords: 1Allergy; 2 Neuromuscular blockers
MeSH Terms: conditions — Hypersensitivity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Blood simple — Single Blood simple at Day 1

SUMMARY:
To assess diagnostic accuracy of flow cytometry applied to the diagnosis of allergy to neuro-muscular blockers and to the determination of the neuro-muscular blocker (NMB) which may be used for an ulterior anaesthesia in case of allergy to one given NMB.

DETAILED DESCRIPTION:
The flow cytometric protocol used for this study, was based on basophil selection by an anti- CCR3 and the analysis of basophil activation by the respective up and down regulation of the CD63 and IgE markers as described previously. Basophil activation was expressed in percentage CD63 expression on activated basophils and in activation index involving IgE and CD63 markers and calculated by a specific algorithm developed by our group.. Our aim is to test a sufficient number of patients in order to be able to establish the ROC curves related to the allergen type tested and validate the use of an allergen mixture (NMB mix containing the 7 usual NMB at the optimal activation concentrations). Patients will be included during the post-anaesthetic consultation on the basis of the diagnosis of an IgE dependant per-anaesthetic reaction. The allegro-anaesthetist diagnostical habits won't be changed.

ELIGIBILITY:
Inclusion Criteria:

* patients aged at least 18 years,
* patients having experienced an IgE dependant per-anaesthetic reaction
* affiliated to a social security

Exclusion criteria:

* patients having taken anti-histamine drugs and corticoids during the last 8 days
* patients submitted to a juridical protection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 129 (Actual)
Dates: Start 2011-04 (Actual); Primary Completion 2019-01 (Actual); Study Completion 2021-01 (Actual)

PRIMARY OUTCOMES:
Allergy diagnosis assessed by cytometry flow data | At Day 1

CONTACTS AND LOCATIONS:
Locations (4):
- France (4):
  - Service d'Allergologie, Angers
  - Service d'Immuno-allergologie, Bordeaux
  - Laboratoire Immunologie et Immunogénétique, Limoges
  - Service d'Anesthésie Réanimation, Nancy

REFERENCES:
- [Background] Place of the basophil activation test in the diagnosis of neuromuscular blocking agent's allergy. Immunological multicenter study